CLINICAL TRIAL: NCT03288272
Title: Evaluation of Repeated Whole Brain Radiotherapy Versus Best Supportive Care for Multiple Brain Metastases - the Randomized Trial ERASER.
Brief Title: Evaluation of Repeated Whole Brain Radiotherapy Versus Best Supportive Care for Multiple Brain Metastases.
Acronym: ERASER
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stephanie Combs (Other)
Responsible Party: Sponsor-Investigator, Stephanie Combs, Professor and Chair, Technical University of Munich
Organization: Technical University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERASER
Record Dates: First submitted 2016-05-15; First posted 2017-09-20 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Brain Metastasases

STUDY DESIGN:
Intervention Model Description: Randomization Best Supportive Care, Two Radiotherapy Dosing Regimens
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 - WBRT 10 x 2 Gy (Active Comparator): Arm 1 - WBRT 10 x 2 Gy Whole brain radiotherapy with a total dose of 20 Gy in single fractions of 2 Gy
  Interventions: Radiation: Whole Brain Radiotherapy
- Arm 2 - WBRT 15 x 2 Gy (Active Comparator): Arm 2 - WBRT 15 x 2 Gy Whole brain radiotherapy with a total dose of 30 Gy in single fractions of 2 Gy
  Interventions: Radiation: Whole Brain Radiotherapy
- Arm 3 - Best Supportive Care (Active Comparator): Symptomatic treatment includes steroids, pain medication, nutritional support etc.
  Interventions: Other: Best Supportive Care

INTERVENTIONS:
Radiation: Whole Brain Radiotherapy — Radiotherapy of the whole brain
  Arms: Arm 1 - WBRT 10 x 2 Gy; Arm 2 - WBRT 15 x 2 Gy
Other: Best Supportive Care — Best Supportive Care including nutrition, pain medication, steroids as needed
  Arms: Arm 3 - Best Supportive Care

SUMMARY:
Whole Brain Radiotherapy (WBRT) has been established as the treatment standard in patients with multiple cerebral metastases from solid tumors. However, intracerebral recurrence is possible and a repeated WBRT may be indicated to improve intracerebral tumor control. Each institutsion offers different dosing regimens, which have all been published to be safe and effective. Some favor best supportive care only.

The current study protocol is aimed at evaluating primarily the toxicity as well as secondarily the local and loco-regional tumor control, overall survival and QoL after repeated WBRT using 2 different dose concepts (20 Gy in 10 Fx vs. 30 Gy in 15 Fx) compared to BSC.

DETAILED DESCRIPTION:
According to Nussbaum et al., 24-45% of cancer patients develop cerebral metastases during the course of the disease. Brain metastases are generally associated with a poor prognosis and high morbidity. Published median survival rates after WBRT are between 2 and 7 months. Standard of care in multiple BM is WBRT delivered as 30 Gy in 10 fractions, leading to modest palliation with a median survival of 3 to 5 months. Prognostic factors include the RPA-classification, performance status, response to steroids and evidence of systemic disease.

Unfortunately, intracerebral recurrence happens. For example, in the cohort of Meyners et al.(2010) on WBRT in relatively radioresistant tumors, median time to recurrence was 4.5months and the local control rates at 6 and 12 months post radiationem were 37% and 15%, respectively. Furthermore, the treatment of intracerebral recurrence after previous WBRT is challenging. In case of </= 3 recurrent BM, surgery or radiosurgery (RS) are options. One other option, especially in case of >3 recurrent BM is repeated WBRT. In this setting, one of the first reports on repeated WBRT was published by Cooper et al. in 1990. The authors reported on repeated WBRT (n=52) consisting of 25 Gy in 10 fractions. Response to reirradiation was seen in 42% of the patients. Furthermore, the patients improved by at least one level in their neurologic function status. Survival after second therapy averaged 5 months. In the report by Wong et al. (1996) median dose of retreatment (n=86) was 20 Gy. Resolution of symptoms was achieved in 27% of patients, partial improvement in 43% and no improvement or worsening of symptoms was seen in 29% of patients. The majority of patients had no significant toxicity secondary to re-irradiation. Five patients had radiographic abnormalities of their brain consistent with radiation-related changes. One patient had symptoms of dementia that was thought to be caused by radiotherapy. Sadikov et al. (2007) reported on 72 patients who underwent repeated WBRT for recurrent or progressive BM. The median survival after re-irradiation was 4.1 months. One patient was reported as having memory impairment and pituitary insufficiency after 5 months of progression-free survival.

In the report by Mayer et al. on re-irradiation tolerance of the human brain -in this analysis focused on recurrent glioma-, the authors concluded that radiation-induced brain tissue necrosis is found to occur at normalized tolerance doses of cumulative > 100 Gy.

The current study protocol is aimed at evaluating primarily the toxicity as well as secondarily the local and loco-regional tumor control, overall survival and QoL after repeated WBRT using 2 different dose concepts (20 Gy in 10 Fx vs. 30 Gy in 15 Fx) compared to BSC.

In the present trial, the primary endpoint toxicity as well as the secondary endpoints QoL, loco-regional progression-free survival, overall survival and imaging response in patients previously treated with WBRT requiring repeated WBRT for intracerebral tumor progression will be evaluated.

ELIGIBILITY:
Inclusion criteria:

* histologically confirmed malignancy
* previous WBRT
* MR-imaging confirmed cerebral metastases (>1)
* age ≥ 18 years of age
* Karnofsky Performance Score ³60
* For women with childbearing potential, (and men) adequate contraception.
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria

* refusal of the patients to take part in the study
* Patients who have not yet recovered from acute high-grade toxicities of prior therapies
* Pregnant or lactating women
* Participation in another clinical study or observation period of competing trials, respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Toxicity | 3 months
  The primary endpoint is toxicity according to CTCAE after whole brain radiotherapy.

SECONDARY OUTCOMES:
loco-regional progression-free survival | 6 months
  follow-up and local control of brain metastases as well as loco-regional control
Quality of Life (QOL) | 6 months
  QOL
Survival | 6 months
  survival after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie E Combs, Prof. Dr., Principal Investigator — Professor and Department Chair
Locations (1):
- Technische Universität München (TUM), Klinikum rechts der Isar, Munich, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Scharp M, Hauswald H, Bischof M, Debus J, Combs SE. Re-irradiation in the treatment of patients with cerebral metastases of solid tumors: retrospective analysis. Radiat Oncol. 2014 Jan 3;9:4. doi: 10.1186/1748-717X-9-4. PMID 24387239